CLINICAL TRIAL: NCT05116709
Title: A Multicenter, Open Phase I Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetic Characteristics and Preliminary Clinical Efficacy of Anti-Tigitmab BAT6005 Injection in Patients with Advanced Malignant Solid Tumors
Brief Title: Assessment of Safety and Preliminary Clinical Efficacy with BAT6005 in Advanced Malignant Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bio-Thera Solutions (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BAT-6005-001-CR
Record Dates: First submitted 2021-10-28; First posted 2021-11-11 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Locally Advanced or Metastatic Solid Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- BAT6005 single drug dose escalation study (Experimental): The whole is divided into two phases.The first stage: 10mg group, 30mg group, 100mg group using accelerated titration method to increase the dose.The second stage: 300mg group, 600mg group, 900mg group according to the standard "3+3" rule dose increase study.
  Interventions: Drug: BAT6005 injection

INTERVENTIONS:
Drug: BAT6005 injection — Six dose groups were set up, including 10mg (initial dose) group, 30mg group, 100mg group, 300mg group, 600mg group and 900mg group, respectively.

SUMMARY:
This research design for center, increasing openness, dose and dose extension phase I clinical trials, research the main evaluation BAT6005 injection single drug in patients with advanced malignant solid tumors in the safety, tolerability and PK characteristics, to explore the maximum tolerated dose and preliminary antitumor efficacy, provide the basis for subsequent clinical trials recommended dose.

Part I: single drug dose escalation study. Part TWO: dose extension study.

DETAILED DESCRIPTION:
The study is divided into two parts:

Part I: single drug dose escalation study. Accelerated titration and "3+3" dose escalation rule were used to explore the safety, tolerability and pharmacokinetic characteristics of BAT6005.

Since the clinical benefit of a single agent may be limited, the study used accelerated titration and the "3+3" dose-escalation rule to explore the safe dose range from the ethical point of view of exposing fewer subjects to ineffective doses.

Six dose groups were set up, including 10mg (initial dose) group, 30mg group, 100mg group, 300mg group, 600mg group and 900mg group, respectively.

The whole is divided into two phases. The first stage: 10mg group, 30mg group, 100mg group using accelerated titration method to increase the dose.

The second stage: 300mg group, 600mg group, 900mg group according to the standard "3+3" rule dose increase study.

Group/Increasing Method Dose group (mg) Number of fixed dose cases (person) A/ Accelerated titration 10 1, or 3~6 B/ Accelerated titration 30 1, or 3~6 C/ accelerated titration 100 1, or 3~6 D/ Standard 3+3 300 3 to 6 E/ Standard 3+3 600 3 to 6 F/ Standard 3+3 900 3 to 6 Note: After the dose-increasing study is completed, it can be considered as appropriate after comprehensive evaluation of safety and other factors, or a new dose can be selected between the dose that stops climbing and the previous lower dose group according to the above rules to determine the more accurate maximum tolerated dose according to the specific situation and the discussion with the researcher.

The dose escalation rules are as follows:

For the first 3 dose groups A, B and C, accelerated titration was used in dose-increasing scheme, i.e. cohort size =1.

First, 1 subject in group A was included. If no grade ≥2 toxicity was observed related to the study drug (except for simple laboratory abnormalities that the investigator judged to be asymptomatic and without intervention), the subject could be directly transferred to group B for dose escalation, which was accelerated to group C by the rule (" 1+1 ").

The accelerated titration dose increase should be discontinued once a class 2 or greater toxicity associated with the drug under study is observed in one group (except for simple laboratory abnormalities that the investigator judged to be asymptomatic and without intervention).

An additional 2 subjects in the dose group will be transferred to the standard "3+3" dose escalation (i.e. cohort size =3) mode until MTD or MAD is reached.

Starting from group D, the dose increasing mode was adjusted to the standard "3+3" rule, as shown in the following table:

DLT population/current dose group population dose increase or decrease decision appears 0/3 3 new subjects received the next high-dose group 1/3 of the current dose group followed by 3 new subjects 1/3 and 0/3 new subjects received the next high-dose group

≥2/3 or ≥2/6 indicates that the dose has exceeded MTD and should be stopped. If there are 6 people in the former dose group, the former lower dose group is used as MTD.

If there are only 3 people in the previous dose group, add 3 people to the previous dose group.

After the addition of 3 persons, MTD continued to be down-regulated if there were ≥2 DLT in the previous dose group If MTD is found, the sponsor may select a dose of MTD or lower as the recommended dose for phase II clinical studies after discussion with the investigator based on the specific situation.

If MTD is not reached, the sponsor may select a dose of MAD or one of the following dose groups as the recommended dose for phase II clinical studies, depending on the specific situation and discussion with the investigator.

As the study progresses, protocols may be allowed to revise the definition of DLT as appropriate in light of new clinical findings.

Adverse events that meet DLT criteria occurring outside the DLT evaluation period or other adverse safety information that the investigator considers meaningful do not directly influence dose-escalation decisions, but should be taken into account in the final determination of THE RP2D.

Prior to each dose increase, the sponsor and investigator will discuss and comprehensively evaluate the decision to increase or decrease the dose, using available information on safety, PK (if any), and efficacy.

Prior to inclusion in the next dose team, all subjects in the previous dose group must complete 21 days of DLT observation before toleration is explored according to the standard "3+3" dose escalation rule.

In dose-escalation studies, the first subject in the same dose group may be included in the next subject 1 week after the first dose observation.

Within each dose group, a minimum of 24 hours should be allowed between the administration of the prior subject and the administration of subsequent subjects.

Dose reduction adjustments are not allowed; The dose of BAT6005 should be upregulated as appropriate, but with extreme caution, at least simultaneously: ① Subjects have received at least 4 cycles of study medication; ② After discussion between the sponsor and the study, it was concluded that the subjects receiving the higher primary dose group might bring more clinical benefits than the current dose group;

③ The higher dose group has been shown to fail to reach MTD by subsequent dose escalation studies.

Part TWO: dose extension study. According to the preliminary safety and efficacy results of the dose-escalation study, the investigator discussed with the sponsor to select the appropriate dose and tumor species for the extended study, so as to further study the safety and clinical efficacy of BAT6005 single drug, providing a basis for subsequent clinical studies.

1~2 dose cohort studies were planned, with no less than 6 patients in each dose cohort, and PK study was carried out.

The overall study period can be roughly divided into screening period, treatment period and follow-up period:

Screening period: -28d~0d, that is, after the informed consent is signed, the screening evaluation can be completed within 28 days.

Treatment period: Every 3 weeks is one administration cycle, the study drug is given on the first day of each cycle, starting from the second cycle, the time window of administration can be ±3 days, but in addition to imaging examination, subjects must complete vital signs, laboratory examination, physical status score and other tests within 3 days before each administration.

Subjects will also be required to complete clinical tumor radiographic evaluations (consistent, CT or MRI) every 6 weeks (±7 days) during the first 24 weeks after initial dosing, and every 9 weeks (±7 days) thereafter.

Study drug therapy should continue until the onset of disease progression, withdrawal due to unacceptable toxicity, acceptance of new antitumor therapy due to lack of therapeutic benefit, withdrawal of informed consent and voluntary withdrawal for other reasons, or a maximum of 17 cycles (approximately 1 year), whichever comes first.

The DLT evaluation period was defined as the first treatment cycle, from initial dosing to 21 days after dosing.

Follow-up Period: If subjects discontinue study drug Therapy, EOT will be considered as the End of Therapy.

All subjects, including those who have discontinued treatment for any reason (except loss of follow-up, death, withdrawal of informed consent), will be scheduled for an EOT visit within 21+7 days of receiving their last study drug or prior to receiving subsequent new antitumor therapy.

EOT visits should include vital signs, physical examination, laboratory examination, and clinical tumor imaging evaluation (CT or MRI).

Safety follow-up:

After receiving the last dose of the study drug, subjects were required to be followed up for safety, including immune-related adverse events (irAE), at 21+7, 60 (±7) days, and 90 (±7) days until 90 (±7) days or after receiving new antitumor therapy.

Safety visits should be conducted at the study center, where vital signs, physical examination, laboratory examination and other examinations should be performed to evaluate AE, concomitant medication and concomitant treatment until the adverse reactions related to the study drug disappear (or reduce to ≤1).

If adverse reactions persist after discontinuation of treatment, the investigator has the discretion to determine the frequency of follow-up based on clinical practice until the investigator believes that the adverse reactions will return to normal, stabilize at an acceptable level, or show no further improvement.

Follow-up for survival: After the safe follow-up, the subjects were followed up once every 12 weeks (±14 days) by telephone until death, loss of follow-up, withdrawal of informed consent or termination of the study.

The longest treatment time of the drugs studied in this project is about 1 year.

If there is no disease progression or intolerance of toxicity after 1 year of initial study use, subjects may return to the study facility for continued use by the investigator.

ELIGIBILITY:
Inclusion Criteria:

1. Age: ≥18 years old, gender: male or female;
2. The expected survival was assessed as at least 3 months;
3. ECOG (Eastern Oncology Collaboration group) physical status score requirement: 0 or 1;
4. Patients with locally advanced or metastatic malignant solid tumors confirmed by histology or cytology without standard therapy, failure of standard therapy, or inapplicable standard therapy;
5. According to RECIST 1.1, there must be evaluable tumor focus in dose increase stage, and at least one measurable tumor focus in dose expansion stage;
6. Fertile women must have a negative serum pregnancy test within 7 days prior to the first dose and be willing to use an effective method of birth control/contraception to prevent pregnancy during the study period up to 6 months after the last dose.Male patients must agree to use an effective contraceptive method for the duration of the study until 6 months after the study's last dosing;Postmenopausal women must be amenorrhea for at least 12 months before they are considered infertile;

Exclusion Criteria:

1. Prior treatment with anti-TiGit monoclonal antibody or anti-TiGit active double antibody;
2. Had received chemotherapy, radiotherapy, biotherapy, endocrine therapy, immunotherapy and other anti-tumor treatments within 4 weeks prior to the first use of the study drug
3. Received other unmarketed investigational drugs or treatments within 4 weeks prior to the first use of the investigational drug;
4. Received live/attenuated vaccine and mRNA vaccine within 4 weeks prior to screening or plan to receive live/attenuated vaccine and mRNA vaccine during the study period;
5. Pregnant or lactating women;
6. Patients whose AE caused by previous anti-tumor therapy did not recover to CTCAE 5.0≤ 1;
7. Patients with cerebral parenchymal metastasis or meningeal metastasis with clinical symptoms, judged by the investigator to be unsuitable for inclusion;
8. Patients who underwent major organ surgery (excluding needle biopsy) or significant trauma within 4 weeks prior to the first use of the study drug, or who required elective surgery during the study period;
9. Those with a history of tissue or organ transplantation;
10. Patients with active infection prior to the first administration and currently requiring intravenous anti-infection therapy;
11. Known history of human immunodeficiency virus (HIV) infection;
12. active hepatitis B;
13. Active HCV infected subjects
14. Subjects with untreated or undergoing treatment for tuberculosis, including but not limited to tuberculosis; Patients who have been prescribed anti-tuberculosis therapy and confirmed by the investigator to have been cured may be included;
15. The subject is known to have a history of severe allergy, or is known to have experienced grade ≥3 allergic reactions to macromolecular protein preparations/monoclonal antibodies in the past;
16. Patients who have active autoimmune diseases, or have had autoimmune diseases with recurrence risk (such as systemic lupus erythematosus, rheumatoid arthritis, vasculitis, etc.), except patients with clinically stable autoimmune thyroid diseases and type I diabetes;
17. Received systemic glucocorticoid (prednisone > 10mg/ day or equivalent dose of the same drug) or other immunosuppressant treatment within 14 days prior to first use of the study drug; The exceptions are local, ocular, intraarticular, intranasal, and inhaled glucocorticoid therapy and short-term prophylaxis (e.g., to prevent contrast agent allergies).
18. IrAE ≥3 has been seen in the past;
19. existing interstitial lung disease;
20. Have a history of serious cardiovascular and cerebrovascular diseases;
21. Third interstitial effusion that could not be controlled clinically was judged not suitable for inclusion by the researcher;
22. Patients with a known history of psychotropic drug abuse or drug use that is considered to affect the compliance of this study;
23. Patients considered unsuitable for the study by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2021-11-12 (Actual); Primary Completion 2024-01-10 (Actual); Study Completion 2024-09-23 (Actual)

PRIMARY OUTCOMES:
Dose-limiting toxicity(DLT) | Complete the first cycle in 21 days
  AE that occur during the dose-limiting toxicity observation period and are considered to be at least possibly related to the drug under study.
Maximum Tolerated dose (MTD) | Complete the first cycle in 21 days
  The highest dose level of DLT observed in ≤1/6 subjects in a dose group during the DLT evaluation period.

SECONDARY OUTCOMES:
Maximum serum drug concentration(Cmax)Pharmacokinetic endpoint | 0-126days
  Pharmacokinetic endpoint
Maximum serum drug time(Tmax) | 0-126days
  Pharmacokinetic endpoint
Half-life period(t1/2)Pharmacokinetic endpoint | 0-126days
  Pharmacokinetic endpoint
Plasma clearance(CL)Pharmacokinetic endpoint | 0-126days
  Pharmacokinetic endpoint
Apparent Volume of Distribution（Vd） | 0-126days
  Pharmacokinetic endpoint
Effect Chamber Elimination Rate Constant（Ke） | 0-126days
  Pharmacokinetic endpoint
Mean Residence Time（MRT） | 0-126days
  Pharmacokinetic endpoint
Area under the curve(AUC0-t, AUC0-inf) | 0-126days
  Pharmacokinetic endpoint
Anti-drug antibodies(ADA)Immunogenic endpoint | 0-126days
  Immunogenicity endpoint
Prevalence of PD-1 receptors on peripheral blood T cells（RO） | 0-126days
  Pharmacodynamics endpoint

OTHER OUTCOMES:
Objective response rate (ORR) | up to 17 cycles（each cycle is 21 days）
  The proportion of patients whose tumors shrink by a certain amount and stay there for a certain amount of time, including CR and PR.
Duration of remission (DOR) | up to 17 cycles（each cycle is 21 days）
  Time from reaching CR or PR to disease progression
Disease control rate (DCR) | up to 17 cycles（each cycle is 21 days）
  Proportion of patients whose tumors shrank or remained stable for a certain amount of time, including CR, PR, and SD
Progression-free survival (PFS) | up to 17 cycles（each cycle is 21 days）
  The time (days) between the date of randomization and the first observation of intracranial or extracranial disease progression (intracranial as determined by imaging or intracranial hypertension, extracranial imaging), and the number of days from the date of randomization to the date of death if the subject died from other causes prior to disease progression.
Overall survival (OS) | up to 17 cycles（each cycle is 21 days）
  From the date of randomization to the time of death from any cause, subjects who were alive at the time of analysis will have their last contact as the cut-off date

CONTACTS AND LOCATIONS:
Overall Officials: Jin Li, Principal Investigator — Shanghai Oriental hospital
Locations (2):
- China (2):
  - Affiliated Cancer Hospital of Shandong First Medical University, Jinan, Shandong
  - Shanghai Oriental hospital, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No